CLINICAL TRIAL: NCT00258804
Title: Evaluation (Safety and Efficacy) of Treatment With Insulin Glargine and Glimepiride in Patients With Type 2 Diabetes Before, During and After the Period of Fasting in Ramadan
Brief Title: Insulin Glargine During and After the Period of Fasting in Ramadan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4055
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
Primary Objectives :

* To compare the number of hypoglycaemic events (severe, symptomatic, asymptomatic, nocturnal) in patients with type 2 diabetes treated with insulin glargine (Lantus®) and glimepiride (Amaryl®), before, during and after the period of fasting in Ramadan.

Secondary Objectives :

* To assess glycaemic control before, during and after Ramadan in terms of HbA1c, FBG, and 8-point blood glucose profile (FBG and 8-point blood glucose profile will be collected with a blood glucose monitor through a monthly patient diary).
* To assess the relationship between hypoglycaemia events during Ramadan and blood glucose control prior and during Ramadan.
* To assess patient satisfaction
* To document adverse events (all serious adverse events, non serious adverse events) throughout the study (all events will be collected through the monthly patient diary).

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria:

* Patients with Type 2 Diabetes mellitus (but without history of ketoacidosis);
* BMI > 25 and < 40 kg/m2;
* Willingness to participate and to fast during Ramadan;
* Patients should be either:

  * Insulin naïve patients
  * Patients already receiving insulin

Exclusion Criteria:

* Pregnancy (as determined by pregnancy blood test at inclusion visit)
* Breast- feeding
* Women of childbearing potential who do not have adequate contraceptive protection
* Need for treatment during the study period with medications that may interfere with the study protocol
* Treatment with any investigational drug (only if in trial) in the last 3 months before entry into the study
* History of drug or alcohol abuse
* Severe and unbalanced diabetic retinopathy
* Clinically relevant cardiovascular, gastrointestinal, hepatic, renal, neurological, endocrine, hematological or other major systemic diseases that may interfere with the study protocol or complicate the interpretation of study results
* Night shift workers

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2005-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Hypoglycaemic events (severe, symptomatic, asymptomatic, nocturnal) before, during and after Ramadan
Glycemic control before, during and after Ramadan in terms of HbA1c, FBG, 8-point blood glucose profile
All other adverse events before, during and after Ramadan
Patient satisfaction before, during and after Ramadan.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick SINNASSAMY, MD, Study Director — Sanofi